CLINICAL TRIAL: NCT04206618
Title: The Role of Myokines in Postmenopausal Osteoporosis
Brief Title: Circulating Myokine Levels and Bone Metabolism
Status: Completed | Type: Observational
Sponsor: 424 General Military Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Athanasios D. Anastasilakis, Principal Investigator, 424 General Military Hospital
Other Study IDs: MYOBONE
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Teriparatide; Denosumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (8):
- premenopausal normal: premenopausal women with normal BMD who will be subjected to a single morning, fasting blood drainage
- postmenopausal normal: postmenopausal women with normal BMD who will be subjected to a single morning, fasting blood drainage
- postmenopausal osteopenia: postmenopausal women with osteopenia who will be subjected to a single morning, fasting blood drainage
- postmenopausal osteoporosis: postmenopausal women with osteoporosis who will be subjected to a single morning, fasting blood drainage
- hip fracture: postmenopausal women at the moment of hip fracture who will be subjected to a single, fasting blood drainage right before osteosynthesis
- controls (knee osteoarthitis): postmenopausal women with knee osteoarthritis who will be subjected to a single, fasting blood drainage right before arthroplasty and serve as controls
- teriparatide group: postmenopausal women with osteoporosis who will be treated with teriparatide (Forsteo) 1 injection of 20mcg subcutaneously daily for 12 months
  Interventions: Drug: Teriparatide
- denosumab group: postmenopausal women with osteoporosis who will be treated with denosumab (Prolia) 1 injection of 60mg subcutaneously every 6 months for 12 months
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Teriparatide — 1 subcutaneous injection daily for 12 months
  Other Names: rhPTH 1-34
  Groups: teriparatide group
Drug: Denosumab — 1 subcutaneous injection every 6 months for 12 months
  Other Names: RANKL inhibitor
  Groups: denosumab group

SUMMARY:
Circulating levels of several myokines will be measured in serum samples obtained from women in various categories of bone density and according to the presence of fracture or not as well as before and after treatment with teriparatide and denosumab

DETAILED DESCRIPTION:
Serum samples for the measurement of several myokines will be obtained from: 1) equal groups of premenopausal women with normal BMD, postmenopausal women with normal BMD, postmenopausal women with osteopenia, and postmenopausal women with osteoporosis; 2) women with hip fracture compared with controls (women subjected to surgery due to knee osteoathritis); 3) women with osteoporosis treated with teriparatide or denosumab for 12 months

ELIGIBILITY:
Inclusion Criteria:

Substudy 1:

• adult women

Substudy 2:

• postmenopausal women with an incident hip fracture

Substudy 3:

• postmenopausal women with osteoporosis

Exclusion Criteria:

* secondary osteoporosis
* any disease that could affect muscle and/or bone metabolism
* any medication that could affect muscle and/or bone metabolism

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women
Study Population: Substudy 1: equal groups (n=25) of premenopausal women with normal BMD, postmenopausal women with normal BMD, postmenopausal women with osteopenia, and postmenopausal women with osteoporosis Substudy 2: postmenopausal women with an incident hip fracture (n=40) compared with controls (postmenopausal women with knee osteoarhtritis) Substudy 3: postmenopausal women with osteoporosis will receive treatment with either teriparatide or denosumab for 12 months
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
follistatin | 0,3,12 months
  circulating levels of myokine follistatin at baseline and their changes at 3 and 12 months with treatment

SECONDARY OUTCOMES:
activin-A | 0,3,12 months
  circulating levels of myokine activin-A at baseline and their changes at 3 and 12 months with treatment
FSTL3 | 0,3,12 months
  circulating levels of myokine FSTL3 at baseline and their changes at 3 and 12 months with treatment
activin-B | 0,3,12 months
  circulating levels of activin-B at baseline and their changes at 3 and 12 months with treatment
irisin | 0,3,12 months
  circulating levels of myokine irisin at baseline and their changes at 3 and 12 months with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Anastasilakis, phD, Principal Investigator — 424 General Military Hospital
Locations (1):
- 424 General Military Hospital, Thessaloniki, Northern Greece, Greece

IPD SHARING:
Plan to Share IPD: Undecided
Data will become available after study completion

REFERENCES:
- [Background] Bowser M, Herberg S, Arounleut P, Shi X, Fulzele S, Hill WD, Isales CM, Hamrick MW. Effects of the activin A-myostatin-follistatin system on aging bone and muscle progenitor cells. Exp Gerontol. 2013 Feb;48(2):290-7. doi: 10.1016/j.exger.2012.11.004. Epub 2012 Nov 21. PMID 23178301
- [Background] Lotinun S, Pearsall RS, Horne WC, Baron R. Activin receptor signaling: a potential therapeutic target for osteoporosis. Curr Mol Pharmacol. 2012 Jun;5(2):195-204. doi: 10.2174/1874467211205020195. PMID 21787285
- [Background] Anastasilakis AD, Polyzos SA, Makras P, Gkiomisi A, Savvides M, Papatheodorou A, Terpos E. Circulating activin-A is elevated in postmenopausal women with low bone mass: the three-month effect of zoledronic acid treatment. Osteoporos Int. 2013 Jul;24(7):2127-32. doi: 10.1007/s00198-012-2198-0. Epub 2012 Nov 3. PMID 23124716
- [Background] Lodberg A, Eijken M, van der Eerden BCJ, Okkels MW, Thomsen JS, Bruel A. A soluble activin type IIA receptor mitigates the loss of femoral neck bone strength and cancellous bone mass in a mouse model of disuse osteopenia. Bone. 2018 May;110:326-334. doi: 10.1016/j.bone.2018.02.026. Epub 2018 Feb 28. PMID 29499419
- [Background] Lotinun S, Pearsall RS, Davies MV, Marvell TH, Monnell TE, Ucran J, Fajardo RJ, Kumar R, Underwood KW, Seehra J, Bouxsein ML, Baron R. A soluble activin receptor Type IIA fusion protein (ACE-011) increases bone mass via a dual anabolic-antiresorptive effect in Cynomolgus monkeys. Bone. 2010 Apr;46(4):1082-8. doi: 10.1016/j.bone.2010.01.370. Epub 2010 Jan 18. PMID 20080223
- [Background] Ruckle J, Jacobs M, Kramer W, Pearsall AE, Kumar R, Underwood KW, Seehra J, Yang Y, Condon CH, Sherman ML. Single-dose, randomized, double-blind, placebo-controlled study of ACE-011 (ActRIIA-IgG1) in postmenopausal women. J Bone Miner Res. 2009 Apr;24(4):744-52. doi: 10.1359/jbmr.081208. PMID 19049340
- [Background] Fahmy-Garcia S, Farrell E, Witte-Bouma J, Robbesom-van den Berge I, Suarez M, Mumcuoglu D, Walles H, Kluijtmans SGJM, van der Eerden BCJ, van Osch GJVM, van Leeuwen JPTM, van Driel M. Follistatin Effects in Migration, Vascularization, and Osteogenesis in vitro and Bone Repair in vivo. Front Bioeng Biotechnol. 2019 Mar 1;7:38. doi: 10.3389/fbioe.2019.00038. eCollection 2019. PMID 30881954
- [Background] Lodberg A, van der Eerden BCJ, Boers-Sijmons B, Thomsen JS, Bruel A, van Leeuwen JPTM, Eijken M. A follistatin-based molecule increases muscle and bone mass without affecting the red blood cell count in mice. FASEB J. 2019 May;33(5):6001-6010. doi: 10.1096/fj.201801969RR. Epub 2019 Feb 13. PMID 30759349
- [Derived] Anastasilakis AD, Polyzos SA, Makras P, Savvidis M, Mantzoros CS. The comparative effect of teriparatide and denosumab on activins, follistatins, and inhibins in women with postmenopausal osteoporosis. J Bone Miner Res. 2024 Sep 2;39(9):1306-1314. doi: 10.1093/jbmr/zjae106. PMID 38976019
- [Derived] Anastasilakis AD, Polyzos SA, Savvidis M, Anastasilakis DA, Sarridimitriou A, Kumar A, Kalra B, Makras P, Mantzoros CS. Association of activins, follistatins and inhibins with incident hip fracture in women with postmenopausal osteoporosis: a proof of concept, case-control study. Endocrine. 2023 Sep;81(3):573-578. doi: 10.1007/s12020-023-03402-x. Epub 2023 May 23. PMID 37221430
- [Derived] Anastasilakis AD, Polyzos SA, Rodopaios NE, Makras P, Kumar A, Kalra B, Mantzoros CS. Activins, follistatins and inhibins in postmenopausal osteoporosis: A proof of concept, case-control study. Metabolism. 2023 Apr;141:155397. doi: 10.1016/j.metabol.2022.155397. Epub 2022 Dec 30. PMID 36587801